CLINICAL TRIAL: NCT03324971
Title: Effect of Reducing Medication Regimen Complexity on Glycemic Control in Patients With Diabetes.
Brief Title: Medication Regimen Complexity and Glycemic Control in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tarek Samy Abdelziz, Senior lecturer, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA-13071
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: A prospective cohort study .The aim of this study to recruit a cohort of diabetic patients,eliminate unnecessary medications,aiming at improving adherence to anti-diabetic medications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetic patients with non-adherence and poly-pharmacy (Experimental): Medications review. Elimination of all unnecessary prescription to cut down the number of medications to the least possible number.
  Interventions: Other: Medications review

INTERVENTIONS:
Other: Medications review — Medications review. Elimination of all unnecessary prescription to cut down the number of medications to the least possible number.
  This is in line with the best practice guidelines.

SUMMARY:
Polypharmacy is an alarming health issue that is defined as prescription of multiple medications, of which some are redundant or unnecessary. Due to comorbidities, diabetic patients are often prescribed multiple medications. Over prescribing occurs either due to, prescribing medications that are not indicated, continuation of certain medications beyond the time of indication, or prescribing more than one medication with the same effect. Improving glycaemic control is the cornerstone for the prevention and treatment of the diabetic complications.

DETAILED DESCRIPTION:
Hypothesis In addition to the side effects and cost of the unnecessary medications, the investigators hypothesis is that poly-pharmacy will adversely affect patients' compliance with the necessary medications.The investigators propose that elimination of unnecessary medications might improve patients' compliance and consequently improve glycemic control diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

All diabetic patients who are eligible by fulfilling all of the following criteria:

1. HGBA1c ≥7 mg/dl.
2. 2) Poly-pharmacy: defined as the use of five or more medications.
3. Non- compliance: patients were surveyed with both direct and indirect methods to identify non adherence.

Exclusion Criteria:

Exclusion after recruitment Any patient whose diabetic medications regimen changed after recruitment due to hospitalisation, illness, stress or patients preference, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | 3 months
  measurement of hemoglobin A1c to determine glycemic control.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek S Abdealziz, Principal Investigator — Cairo University
Locations (1):
- Cairo university hospitals, Cairo, Egypt